CLINICAL TRIAL: NCT00001151
Title: Studies With 1,25-Dihydroxycholecalciferol
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated because of lack of drug supply
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Stephen Marx, M.D., Chief of the Metabolic Diseases Branch of NIDDK/NIH, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 760081; 76-DK-0081 (Other: 76-DK-0081)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-06

CONDITIONS: Hypocalcemia; Rickets
Keywords: Calciferol; Hypocalcemia; Rickets
MeSH Terms: conditions — Hypocalcemia; Rickets | interventions — Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug treatment (Experimental): 1,25-Dihydroxycholecalciferol 5 ug orally per day for 2 years
  Interventions: Drug: 1,25-Dihydroxycholecalciferol

INTERVENTIONS:
Drug: 1,25-Dihydroxycholecalciferol — Usual doses of 1,25-dihydroycholecalciferol are 0.25-1 ug per day. All patients in this study received very high doses or 5-20 ug per day.

SUMMARY:
Vitamin D in the diet undergoes changes in the liver and kidneys to several forms. Patients suffering from disorders with Vitamin D resistance are unable to absorb calcium from food. Patients diagnosed with these disorders will be evaluated and treated with high doses of another form of Vitamin D (1,25-dihydroxyvitamin D3). Patients will be monitored and observed throughout the study to avoid experiencing side effects from the medication.

DETAILED DESCRIPTION:
Patients with extreme resistance to 1,25-dihydroxyvitamin D will be evaluated and treated with high doses of 1,25-dihydroxyvitamin D3.

Plan: In previously untreated patients the study will be divided into a control and one or more treatment periods. During the control period, parathyroid status will be assessed by parameters nos. 1& 2 (below). In previously treated patients maintenance vitamin D will be gradually replaced with 1,25(OH)2D3. This will be accomplished by withdrawal of vitamin D and institution of 1,25(OH)2D3 when the serum calcium shows a downward trend.

1,25(OH)2D3 as 0.25 or 0.5 ug capsules (though IND 20,889) or as a solution of I microgram per ml will be administered orally. In most cases, because of consideration of time and expense, the cooperation of the patient's local physician will be enlisted. The following will be monitored:

1. Serum calcium, phosphorus,alkaline phosphatase,creatinine at twice weekly intervals. After a maintenance dose has been established, this will be decreased to a monthly, and subsequently 3-6 monthly interval.
2. Urine calcium, phosphorus,creatinine and cAMP before therapy and, when appropriate, during therapy.

The dose of 1,25(OH)2D3 will be 0.125 to 50.0 ug/day. Serum calcium will not be allowed to rise above the normal range (2.0 -2.4 mM at NIH). Should hypercalcemia occur, appropriate treatment will be initiated and the drug dosage will be decreased.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with hereditary resistance to calcitrol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 1976-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Marx, MD, Principal Investigator — NIDDK/NIH
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Marx SJ, Swart EG Jr, Hamstra AJ, DeLuca HF. Normal intrauterine development of the fetus of a woman receiving extraordinarily high doses of 1,25-dihydroxyvitamin D3. J Clin Endocrinol Metab. 1980 Nov;51(5):1138-42. doi: 10.1210/jcem-51-5-1138. PMID 6893458
- [Background] Fraser D, Kooh SW, Kind HP, Holick MF, Tanaka Y, DeLuca HF. Pathogenesis of hereditary vitamin-D-dependent rickets. An inborn error of vitamin D metabolism involving defective conversion of 25-hydroxyvitamin D to 1 alpha,25-dihydroxyvitamin D. N Engl J Med. 1973 Oct 18;289(16):817-22. doi: 10.1056/NEJM197310182891601. No abstract available. PMID 4357855
- [Background] Marx SJ, Spiegel AM, Brown EM, Gardner DG, Downs RW Jr, Attie M, Hamstra AJ, DeLuca HF. A familial syndrome of decrease in sensitivity to 1,25-dihydroxyvitamin D. J Clin Endocrinol Metab. 1978 Dec;47(6):1303-10. doi: 10.1210/jcem-47-6-1303. PMID 233695

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Patient has rickets (child) or osteomalacia (adult) of bone
Period: Overall Study
Arm/Group | Group 1
Started | 6
Completed | 1
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Patient has rickets (cild) or osteomalacia (adult) of bone
Arm/Group | Group 1
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 15 [5 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Normal Serum Calcium Concentrations
Description: Normal calcium concentration 8.2-10.6 mg/dL
Time Frame: 1 year average
Measure: Number; unit: participants
Arm/Group | Group 1
Number analyzed (Participants) | 6
participants | 6 [8 to 11]

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes